CLINICAL TRIAL: NCT04645355
Title: Immunogenetic Profiling of Guselkumab for the Treatment of Plaque and Guttate Psoriasis
Brief Title: Guselkumab Immunogenetics
Acronym: TIG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-32273
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis Guttate; Plaque Psoriasis
MeSH Terms: conditions — Guttate Psoriasis | interventions — guselkumab

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label study. Twenty-five subjects are planned (15 with new-onset guttate psoriasis and 10 with chronic plaque psoriasis). Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. All subjects will initially be treated with guselkumab 100 mg SQ at weeks 0, 4, and then every 8 weeks thereafter until week 44.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- New-onset guttate psoriasis (Experimental): Subjects will initially be treated with guselkumab 100 mg SQ at weeks 0, 4, and then every 8 weeks thereafter until week 44. At week 44, patients who have not achieved PASI 50 (nonresponders) will be removed from the trial. Patients who achieve between PASI 50 and PASI 75 (partial responders) will continue on drug throughout the remainder of the study. Patients who achieve PASI 75 or greater at week 44 (responders) will have their guselkumab therapy withdrawn and re-treated upon relapse.
  Interventions: Drug: Guselkumab
- Chronic plaque psoriasis (Experimental): Subjects will initially be treated with guselkumab 100 mg SQ at weeks 0, 4, and then every 8 weeks thereafter until week 44. At week 44, patients who have not achieved PASI 50 (nonresponders) will be removed from the trial. Patients who achieve between PASI 50 and PASI 75 (partial responders) will continue on drug throughout the remainder of the study. Patients who achieve PASI 75 or greater at week 44 (responders) will have their guselkumab therapy withdrawn and re-treated upon relapse.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — All subjects will initially be treated with guselkumab 100 mg SQ at weeks 0, 4, and then every 8 weeks thereafter until week 44

SUMMARY:
This is a two-arm open-label study to evaluate the clinical and immunogenetic responses of patients with plaque or guttate psoriasis to treatment with guselkumab.

DETAILED DESCRIPTION:
Guselkumab (Tremfya®), an IL-23 inhibitor approved for the treatment of moderate-to-severe plaque psoriasis. Given the potential role of IL-23 in the pathogenesis of guttate psoriasis, guselkumab may be an effective option to treat the initial manifestation of guttate psoriasis. This is a two-arm open-label study to evaluate the clinical and immunogenetic responses of patients with plaque or guttate psoriasis to treatment with guselkumab. The primary objective of this study is to assess how treatment with guselkumab changes the immune milieu of the skin in patients with plaque or guttate psoriasis. The secondary objectives of this study are to assess how treatment with guselkumab affects the quality of life and extent of skin disease in patients with plaque or guttate psoriasis.

ELIGIBILITY:
Inclusion Criteria:

For subjects with guttate psoriasis:

* Ability to provide written informed consent and comply with the protocol.
* At least 18 years of age.
* Diagnosis of guttate psoriasis.
* Onset of guttate psoriasis within 12 months.
* Body surface area (BSA) involvement greater than or equal to 5%.
* PASI greater than or equal to 4.
* Subject is considered a candidate for phototherapy or systemic therapy.
* Subject is unlikely to conceive due to male, post-menopausal, or using adequate contraceptive (barrier, hormonal, implant, or permanent sterilization methods). Women of childbearing potential will be allowed to enroll provided they practice adequate forms of birth control.
* Physical exam with no evidence of active skin infection and/or other findings that indicate chronic disease or concomitant inflammatory/immune-mediated skin disease other than psoriasis.

For subjects with chronic plaque psoriasis (control):

* Ability to provide written informed consent and comply with the protocol.
* At least 18 years of age.
* Diagnosis of plaque psoriasis.
* Duration of plaque psoriasis >5 years.
* Body surface area (BSA) involvement greater than or equal to 5%.
* Subject is considered a candidate for phototherapy or systemic therapy.
* Subject is unlikely to conceive due to male, post-menopausal, or using adequate contraceptive (barrier, hormonal, implant, or permanent sterilization methods). Women of childbearing potential will be allowed to enroll provided they practice adequate forms of birth control.
* Physical exam with no evidence of active skin infection and/or other findings that indicate chronic disease or concomitant inflammatory/immune-mediated skin disease other than psoriasis.

Exclusion Criteria:

For subjects with guttate psoriasis:

* Subject is unable to provide written informed consent or comply with the protocol.
* Subject is younger than 18 years of age or older than 70 years.
* Have a history of active, chronic or recurrent infectious disease including HIV, hepatitis B, or hepatitis C.
* Have active tuberculosis or latent tuberculosis without at least 4 weeks of treatment with isoniazid.
* Have current signs or symptoms of severe, progressive, or uncontrolled medical disease.
* Known allergies, hypersensitivity, or intolerance to guselkumab (TremfyaTM) excipients.
* Have a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to screening)
* Are pregnant, nursing, or planning a pregnancy while enrolled in the study or for 12 weeks after the study agent injection for women or are planning to father a child while enrolled in the study or for 12 weeks after the last study agent injection.
* Are participating in another study using an investigational agent or procedure during participation in this study.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.
* Subjects possess other diagnoses that, in the investigator's opinion interfere with the evaluation of the subject's guttate psoriasis.
* Pre-existing psoriasis of any type for longer than 6 months. (i.e. plaque, guttate, palmoplantar, pustular, erythrodermic)
* Previous treatment for psoriasis with phototherapy (narrowband ultraviolet (UV) B, broadband UVB, or UVA), systemic agents (methotrexate, acitretin, cyclosporine, apremilast), or biologic agents (etanercept, adalimumab, ustekinumab, secukinumab, etc.)

For subjects with chronic plaque psoriasis:

* Subject is unable to provide written informed consent or comply with the protocol.
* Subject is younger than 18 years of age or older than 70 years.
* Have a history of active, chronic or recurrent infectious disease, including HIV, hepatitis B, or hepatitis C.
* Have active tuberculosis or latent tuberculosis without at least 4 weeks of treatment with isoniazid.
* Have current signs or symptoms of severe, progressive, or uncontrolled medical disease.
* Known allergies, hypersensitivity, or intolerance to guselkumab (TremfyaTM) excipients.
* Have a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to screening)
* Are pregnant, nursing, or planning a pregnancy while enrolled in the study or for 12 weeks after the study agent injection for women or are planning to father a child while enrolled in the study or for 12 weeks after the last study agent injection.
* Are participating in another study using an investigational agent or procedure during participation in this study.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.
* Subjects possess other diagnoses that, in the investigator's opinion, interfere with the evaluation of the subject's plaque psoriasis.
* Prior history of guttate psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Lesional CD4+ T effector cells | baseline and week 44
  Mean change from baseline in percent of lesional CD4+ T effector cells producing IL-17
Lesional CD8+ T effector cells | baseline and week 44
  Mean change from baseline in percent of lesional CD8+ T effector cells producing IL-17

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Liao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Non-identifying clinical and research data may be shared with Janssen Biotech, UCSF and FDA, as well as other qualified scientists upon publication and upon request